CLINICAL TRIAL: NCT03807739
Title: A Phase I Study to Determine the Relative Bioavailability of Various Formulations of GDC-0134 in Healthy Female Subjects of Non-Childbearing Potential
Brief Title: A Study to Determine the Bioavailability of Various Formulations of GDC-0134 in Healthy Female Participants of Non-Childbearing Potential
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: GP40957
Record Dates: First submitted 2019-01-15; First posted 2019-01-17 (Actual); Results first posted 2020-08-31 (Actual); Last update posted 2020-08-31 (Actual); Status verified 2020-08

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part I: GDC-0134 F16 vs F09 Capsule Formulation (Experimental): In Part 1 participants will receive single doses of either GDC-0134 F16 capsules (prototype) or GDC-0134 F09 capsules (reference) after having consumed a standard meal.
  Interventions: Drug: GDC-0134 F09 Formulation; Drug: GDC-0134 F16 Formulation
- Part II: GDC-0134 F15 vs F09 Capsule Formulation (Experimental): In Part 2, participants will receive a single dose of either GDC-0134 F15 capsules (prototype) or GDC-0134 F09 capsules (reference) after an overnight fast.
  Interventions: Drug: GDC-0134 F09 Formulation; Drug: GDC-0134 F15 Formulation

INTERVENTIONS:
Drug: GDC-0134 F09 Formulation — Participants will receive a single oral dose of GDC-0134 reference capsule F09.
Drug: GDC-0134 F15 Formulation — Participants will receive a single oral dose of GDC-0134 prototype capsule F15.
  Arms: Part II: GDC-0134 F15 vs F09 Capsule Formulation
Drug: GDC-0134 F16 Formulation — Participants will receive a single oral dose of GDC-0134 prototype capsule F16.
  Arms: Part I: GDC-0134 F16 vs F09 Capsule Formulation

SUMMARY:
This is a two-part study to determine the relative bioavailability of two different prototype capsules of GDC-0134 to that of an existing reference capsule of GDC-0134 under both fed and fasted conditions. The study is open to healthy female participants of non-childbearing potential.

ELIGIBILITY:
Inclusion Criteria

* Body mass index (BMI) range 18.5 to 35 kilograms per square meter (kg/m2)
* In good health, determined by no clinically significant findings from medical history, physical examination, 12-lead ECG, and vital signs;
* Clinical laboratory evaluations within the reference range for the test laboratory, unless deemed not clinically significant by the principal investigators (PIs)
* Females of non-childbearing potential only

Exclusion Criteria

* History or clinical manifestation of any significant medical condition as determined by the PI (or designee)
* History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the PI (or designee)
* History of stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs
* Use of any prescription medications/products within 14 days prior to Check-in (Day -1) for their first treatment period and during the entire study duration, unless deemed acceptable by the PI
* Use of oral antibiotics within 4 weeks or intravenous antibiotics within 8 weeks prior to the Screening evaluation and during the entire study duration
* Use of any over-the-counter, non-prescription preparations within 14 days prior to Check-in (Day -1) for their first treatment period and during the entire study duration, unless deemed acceptable by the PI
* Use of acid reducing medications (proton pump inhibitors [PPIs], histamine H2-receptor antagonists [H2RAs]) within 14 days prior to Check-in (Day -1) for their first treatment period and during the entire study duration. As an alternative, antacids may be allowed at least 4 hours before or after dose
* Use of any vaccines (including seasonal flu and H1N1 vaccines) within 14 days prior to Check-in (Day -1) for their first treatment period
* Use of tobacco- or nicotine-containing products within 6 months prior to Check-in (Day -1) for their first treatment period and during the entire study
* Any acute or chronic condition or any other reason that, in the opinion of the PI, would limit the subject's ability to complete and/or participate in this clinical study

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Healthy female participants of non-childbearing potential
Enrollment: 38 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2019-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (2):
- United States (2):
  - Covance Research Unit - Daytona, Daytona Beach, Florida
  - Covance Research Unit - Dallas, Dallas, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Screening period: Day -28 to Day 2
Groups:
- Part 1: GDC-0134 F09 vs GDC-0134 F16 Capsule Formulation: In Part 1 participants received single doses of either GDC-0134 F09 or GDC-0134 F16 capsules (prototype) after having consumed a standard meal.
- Part 1: GDC-0134 F16 vs GDC-0134 F09 Capsule Formulation: In Part 1, participants received a single dose of either GDC-0134 F16 capsules or GDC-0134 F09 capsules after after having consumed a standard meal.
- Part 2: GDC-0134 F09 vs GDC-0134 F15 Capsule Formulation: In Part 2 participants received single doses of either GDC-0134 F09 or GDC-0134 F15 capsules (prototype) in fasting conditions.
- Part 2: GDC-0134 F15 vs GDC-0134 F09 Capsule Formulation: In Part 2 participants received single doses of either GDC-0134 F15 or GDC-0134 F09 capsules (prototype) in fasting conditions.
Period: Overall Study
Arm/Group | Part 1: GDC-0134 F09 vs GDC-0134 F16 Capsule Formulation | Part 1: GDC-0134 F16 vs GDC-0134 F09 Capsule Formulation | Part 2: GDC-0134 F09 vs GDC-0134 F15 Capsule Formulation | Part 2: GDC-0134 F15 vs GDC-0134 F09 Capsule Formulation
Started | 9 | 10 | 9 | 10
Completed | 7 | 10 | 9 | 10
Not Completed | 2 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Part I: GDC-0134 F09 vs GDC-0134 F16 Capsule Formulation: In Part 1 participants received single doses of either GDC-0134 F09 capsules (prototype) or GDC-0134 F16 capsules (reference) after having consumed a standard meal.
- Total: Total of all reporting groups
Arm/Group | Part I: GDC-0134 F09 vs GDC-0134 F16 Capsule Formulation | Part 1: GDC-0134 F16 vs GDC-0134 F09 Capsule Formulation | Part 2: GDC-0134 F09 vs GDC-0134 F15 Capsule Formulation | Part 2: GDC-0134 F15 vs GDC-0134 F09 Capsule Formulation | Total
Number analyzed (Participants) | 9 | 10 | 9 | 10 | 38
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.3 (8.9) | 56.5 (4.8) | 52.6 (7.2) | 58.8 (3.1) | 56.1 (6.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 9 | 10 | 38
  Male | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 3 | 4 | 12
  Not Hispanic or Latino | 6 | 8 | 6 | 6 | 26
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 3 | 2 | 2 | 8
  White | 8 | 7 | 7 | 8 | 30
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Weight [Mean (Standard Deviation); unit: kg] | 74.5 (12.5) | 68.9 (10.9) | 73.4 (15.6) | 71.5 (10.0) | 72.0 (12.0)
Height [Mean (Standard Deviation); unit: cm] | 162.9 (7.6) | 161.2 (5.8) | 159.1 (6.6) | 160.6 (5.0) | 160.9 (6.2)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 28.1 (4.2) | 26.7 (5.0) | 159.1 (4.4) | 27.9 (5.1) | 27.8 (4.6)

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Concentration (Cmax) of GDC-0134.
Time Frame: The time points at which the outcome measure was assessed were 0, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 96, 144, 336, 504 hours post-dose.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: uM
Groups:
- Part 1 GDC-0134 F16 Capsule Fed: In Part 1 participants received single doses of GDC-0134 F16 after having consumed a standard meal.
- Part 1 GDC-0134 F09 Capsule Fed: In Part I participants received single doses of GDC-0134 F09 capsules after having consumed a standard meal.
- Part 2 GDC-0134 F15 Fasted: In Part 2, participants received a single dose of GDC-0134 F15 capsules after an overnight fast.
- Part 2 GDC-0134 F09 Capsule Fasted: In Part 2, participants received a single dose of GDC-0134 F09 capsules after an overnight fast.
Arm/Group | Part 1 GDC-0134 F16 Capsule Fed | Part 1 GDC-0134 F09 Capsule Fed | Part 2 GDC-0134 F15 Fasted | Part 2 GDC-0134 F09 Capsule Fasted
Number analyzed (Participants) | 18 | 19 | 19 | 19
uM | 5.56 (85.2) | 4.45 (93.7) | 2.66 (131.5) | 2.68 (140.1)
Statistical Analysis 1: Comparison: Part 1 GDC-0134 F16 Capsule Fed vs Part 1 GDC-0134 F09 Capsule Fed; Test type: Equivalence — Equivalence margin 80% - 125%; Geometric LS Mean Ratio = 1.2471, 90% CI 2-sided [1.1149 to 1.3951]
Statistical Analysis 2: Comparison: Part 2 GDC-0134 F15 Fasted vs Part 2 GDC-0134 F09 Capsule Fasted; Test type: Equivalence — Equivalence margin 80% - 125%; Geometric LS Mean Ratio = 0.9864, 90% CI 2-sided [0.8531 to 1.1405]

2. Secondary Outcome: Percentage of Participants With Adverse Events (AEs)
Time Frame: From baseline through the end of study (approximately 11 weeks)
Measure: Number; unit: Percentage of Participants
Groups:
- Part II: GDC-0134 F15 vs F09 Capsule Formulation: In Part 2, participants received a single dose of either GDC-0134 F15 capsules (prototype) or GDC-0134 F09 capsules (reference) after an overnight fast.
Arm/Group | Part I: GDC-0134 F09 vs GDC-0134 F16 Capsule Formulation | Part II: GDC-0134 F15 vs F09 Capsule Formulation
Number analyzed (Participants) | 19 | 19
Percentage of Participants | 63.2 | 52.6

3. Primary Outcome: Area Under the Curve Extrapolated to Infinity (AUCinf) of GDC-0134
Time Frame: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: uM.h
Arm/Group | Part 1 GDC-0134 F16 Capsule Fed | Part 1 GDC-0134 F09 Capsule Fed | Part 2 GDC-0134 F15 Fasted | Part 2 GDC-0134 F09 Capsule Fasted
Number analyzed (Participants) | 18 | 19 | 19 | 19
uM.h | 190 (78.7) | 154 (94.9) | 84.8 (103.4) | 85.6 (103.9)
Statistical Analysis 1: Comparison: Part 1 GDC-0134 F16 Capsule Fed vs Part 1 GDC-0134 F09 Capsule Fed; Test type: Equivalence — Equivalence margin 80% - 125%; Geometric LS Mean Ratio = 1.2203, 90% CI 2-sided [1.1175 to 1.3327]
Statistical Analysis 2: Comparison: Part 2 GDC-0134 F15 Fasted vs Part 2 GDC-0134 F09 Capsule Fasted; Test type: Equivalence — Equivalence margin 80% - 125%; Geometric LS Mean Ratio = 0.9947, 90% CI 2-sided [0.8266 to 1.1968]

ADVERSE EVENTS:
Time Frame: From baseline up to 4 months
Description: The pre-specified intent of the study was to assess the adverse events in participants receiving GDC-0134, regardless of which formulation was given (e.g., F09 vs F16), therefore, all participants receiving GDC-0134 are combined into a single Arm, for each part.
Arm/Group | Part I: GDC-0134 F09 vs GDC-0134 F16 Capsule Formulation | Part II: GDC-0134 F15 vs F09 Capsule Formulation
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 10/19 | 10/19
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part I: GDC-0134 F09 vs GDC-0134 F16 Capsule Formulation (N=19) | Part II: GDC-0134 F15 vs F09 Capsule Formulation (N=19)
Headache (Nervous system disorders) | 7 (9) | 7 (8)
Dizziness (Nervous system disorders) | 1 (1) | 3 (3)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (2) | 4 (5)
Vomiting (Gastrointestinal disorders) | 1 (1) | 4 (4)
Haemoglobin decreased (Investigations) | 2 (4) | 0 (0)
Haematocrit decreased (Investigations) | 1 (1) | 0 (0)
Mean cell volume decreased (Investigations) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Vessel puncture site swelling (General disorders) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 3 (3)
Asthenia (General disorders) | 0 (0) | 1 (1)
Eye pain (Eye disorders) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (1)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2018-12-19): https://cdn.clinicaltrials.gov/large-docs/39/NCT03807739/Prot_000.pdf
  • Statistical Analysis Plan (2019-03-01): https://cdn.clinicaltrials.gov/large-docs/39/NCT03807739/SAP_001.pdf